CLINICAL TRIAL: NCT06949423
Title: Accessing the Impact of Deep TMS Neuromodulation on Neural Circuits Associated With Alcohol Use Disorder
Brief Title: Assessing the Impact of Deep TMS Neuromodulation on Neural Circuits Associated With Alcohol Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Claudia Padula, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 78836; R01AA031552 (NIH)
Record Dates: First submitted 2025-04-07; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder (AUD); Transcranial Magnetic Stimilation
Keywords: Veterans; Deep Transcranial Magnetic Stimulation (dTMS); Neuroimaging; Relapse
MeSH Terms: conditions — Alcoholism; Recurrence

STUDY DESIGN:
Intervention Model Description: 2-arm, 1:1 ratio, randomized, double-blind, sham-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be completed and stored with staff in the Biostatistic Core. Treatment assignments will be recorded on a USB drive read by the device in order to ensure treaters and study investigators remain blinded. In the instance that a serious adverse event (SAE) occur, consultation with the Data Safety and Monitoring Board and the Institutional Review Board will occur to determine the appropriateness of breaking the blind. The blind may be broken for a specific individual in order to determine whether the SAE is related to the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active dTMS (Experimental): Participants will receive 30 sessions of active-dTMS to the dACC/mPFC with the H7 coil, administered 3 times per day over 10 consecutive business days. Each treatment visit will last approximately 30 minutes in total.
  Interventions: Device: Deep Transcranial Magnetic Stimulation (dTMS) H7 coil - Active
- Sham dTMS (Sham Comparator): Participants will receive 30 sham dTMS sessions, administered 3 times per day over 10 consecutive business days. Each treatment visit will last approximately 30 minutes in total.
  Interventions: Device: Deep Transcranial Magnetic Stimulation (dTMS) H7 coil - Sham

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation (dTMS) H7 coil - Active — The study will utilize the H7 coil to administer active Deep Transcranial Magnetic Stimulation (dTMS) to the dorsal anterior cingulate cortex (dACC), a core salience network node.
  Arms: Active dTMS
Device: Deep Transcranial Magnetic Stimulation (dTMS) H7 coil - Sham — The study will utilize an identical protocol using the H7 coil to administer a sham condition.
  Arms: Sham dTMS

SUMMARY:
The purpose of this study is to evaluate the efficacy of deep transcranial magnetic stimulation as a treatment for Veterans with Alcohol Use Disorder (AUD) to decrease the exceedingly high rate of relapse associated with this condition.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is a highly prevalent disorder with a chronic relapse-remit cycle, and over 60% of individuals relapse within months of treatment. Preclinical and human research over the last several decades have defined AUD as a neural circuit-based disorder, which are driven by changes in salience network (SN) function. Emerging non-invasive neuromodulation techniques, such as deep transcranial magnetic stimulation (dTMS), can directly modify neural targets that are related to AUD relapse risk, including the SN.

Preclinical and clinical studies have shown that manipulation of deep cortical nodes within the salience network (SN), such as the dorsal anterior cingulate cortex (dACC), can reduce compulsive drinking. Our lab has demonstrated that blunted dACC activation to affective cues predicts relapse - identifying dACC as a promising neuromodulation target. A systematic interrogation of salience network neuromodulation bridges preclinical and clinical research and has the potential to revolutionize AUD treatment. Our preliminary data demonstrates 1) feasibility of the proposed dTMS protocol and 2) promising neural and clinical outcomes. Specifically, those who received this innovative intervention demonstrated increased dACC activation to affective cues from pre- to post-treatment, dynamic changes in functional connectivity and 100% abstinence at follow up.

Building on these data and a theory-driven conceptual framework, the current proposal aims to systematically address three remaining scientific gaps: 1) to what extent does dTMS stimulation of the dACC modify drinking rates and neural targets, 2) can target engagement be a marker of early treatment response, and 3) how long do the effects of dTMS last? This research is significant and innovative as it utilizes a novel, neuromodulation technique to directly manipulate neural networks that drive relapse in AUD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75.
* Current DSM-5 diagnosis of moderate to severe AUD (≥4 diagnostic symptoms).
* Ability to obtain a Motor Threshold (MT) will be determined during the screening process.
* Has an adequately stable condition and environment to enable attendance at scheduled clinic visits.
* Able to read, understand and voluntarily sign the Informed Consent Form prior to participating in any study-specific procedures or assessments.
* If on a medication regimen for comorbid symptoms, that regimen will be stable for the duration of the study and patient will be willing to remain on this regimen during the treatment phase.
* Fluency in English.

Exclusion Criteria:

* Transcranial magnetic stimulation (TMS) and magnetic resonance imaging (MRI) contraindications: such as a cardiac pacemaker, cochlear implant, or an implanted device (deep brain stimulation, metal in the head, metal in the body, claustrophobia, pregnant or breastfeeding or other ferromagnetic device/objected in the head and body within 30 cm of the treatment coil.
* General medical condition, disease or neurological disorder that interferes with the assessments or participation.
* Unable to safely withdraw, at least two weeks prior to treatment, from medications that increase seizure risk.
* Current substance abuse (except caffeine or nicotine) as determined by positive toxicology screen.
* Have a mass lesion, cerebral infarct, or other active CNS disease, including an alcohol-related seizure or a seizure disorder.
* A recent suicide attempt (defined as within the last 30 days) or presence of current suicidal plan or intent. Patients at risk for suicide will be required to establish a written safety plan involving their primary therapist before entering the study.
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with the ability to follow study protocols.
* Greater than mild traumatic brain injury (defined as greater than 10 minutes loss of consciousness).
* Taking benzodiazepine or neuroleptic medications, or any medication known to alter seizure threshold
* Acute or unstable chronic illness.
* Current or lifetime history of bipolar disorder or psychosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Dorsal Anterior Cingulate Cortex Function (dACC) Activation During the FACES Task, Measured via fMRI | 1-4 days post treatment
  dACC activation to threat faces will be measured using fMRI during the FACES task, designed to assess emotional processing. Activation will be quantified as percent signal change from baseline (pre-treatment) to post-treatment scan.
Percentage of Days Abstinent from Alcohol, Assessed by Timeline Followback (TLFB) | 3-months post treatment
  Alcohol abstinence will be assessed using the TLFB structured interview method. The outcome will be calculated as the percentage of alcohol-free days out of the total number of days in the 3-month follow-up period post-treatment.
Percentage of Heavy Drinking Days, Assessed by Timeline Followback (TLFB) | 3 months post-treatment
  Heavy drinking days are defined as ≥5 drinks/day for men and ≥4 drinks/day for women within a 2-hour period. Self-reported data via TLFB used to calculate the percentage of heavy drinking days during the 3-month follow-up treatment.

SECONDARY OUTCOMES:
Change in Salience Network Functional Connectivity During FACES Task, Measured via fMRI | 1-4 days post treatment
  Functional connectivity between the dACC and prefrontal cortex (PFC) will be assessed using fMRI during the FACES Task. Connectivity strength will be calculated using psychophysiological interaction (PPI) analysis or similar methods.
Change in Resting-State Salience Network Activation, Measured via fMRI | 1-4 days post-treatment
  Resting-state fMRI will assess dACC activation. Measures will include percent signal change pre- to post-treatment.
Change in Resting-State Salience Network Functional Connectivity, Measured via fMRI | 1-4 days post treatment
  Resting-state functional connectivity between the dACC and prefrontal cortex (PFC) will be measured using CONN.
Relapse Status, assessed by Timeline Followback (TLFB) | 3 months post-treatment
  Relapse will be defined as any alcohol use following the post-treatment period, assessed using TLFB. Outcome will be reported as a binary (yes/no) variable.
Total Number of Alcoholic Drinks Consumed, Assessed by Timeline Followback (TLFB) | 3 months post-treatment
  Self-reported alcohol use over the 3-month follow-up period will be assessed via TLFB, and the total number of standard alcoholic drinks consumed will be calculated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia B Padula, PhD, Principal Investigator — Stanford University; Michelle R Madore, PhD, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data, specimens, forms, reports, and other records that leave the site will be identified only by a participant ID number to maintain confidentiality. The ID Number will have no relationship to any aspect of identifiable private information. Therefore, the data associated with each participant will be completely de-identified and there will be no mechanism by which users can re-identify participant data (e.g., name, address) with the subject code.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Three to twelve months after publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Padula CB, Tenekedjieva LT, McCalley DM, Al-Dasouqi H, Hanlon CA, Williams LM, Kozel FA, Knutson B, Durazzo TC, Yesavage JA, Madore MR. Targeting the Salience Network: A Mini-Review on a Novel Neuromodulation Approach for Treating Alcohol Use Disorder. Front Psychiatry. 2022 May 17;13:893833. doi: 10.3389/fpsyt.2022.893833. eCollection 2022. PMID 35656355
- [Background] Padula CB, Tenekedjieva LT, McCalley DM, Morales JM, Madore MR. Accelerated deep TMS in alcohol use disorder: A preliminary pilot trial targeting the dorsal anterior cingulate cortex increases neural target engagement and abstinence. Brain Stimul. 2024 Sep-Oct;17(5):1098-1100. doi: 10.1016/j.brs.2024.09.002. Epub 2024 Sep 13. No abstract available. PMID 39265786
- [Background] Harel M, Perini I, Kampe R, Alyagon U, Shalev H, Besser I, Sommer WH, Heilig M, Zangen A. Repetitive Transcranial Magnetic Stimulation in Alcohol Dependence: A Randomized, Double-Blind, Sham-Controlled Proof-of-Concept Trial Targeting the Medial Prefrontal and Anterior Cingulate Cortices. Biol Psychiatry. 2022 Jun 15;91(12):1061-1069. doi: 10.1016/j.biopsych.2021.11.020. Epub 2021 Dec 6. PMID 35067356
- [Background] Peters SK, Dunlop K, Downar J. Cortico-Striatal-Thalamic Loop Circuits of the Salience Network: A Central Pathway in Psychiatric Disease and Treatment. Front Syst Neurosci. 2016 Dec 27;10:104. doi: 10.3389/fnsys.2016.00104. eCollection 2016. PMID 28082874
- [Background] Koob GF, Volkow ND. Neurocircuitry of addiction. Neuropsychopharmacology. 2010 Jan;35(1):217-38. doi: 10.1038/npp.2009.110. PMID 19710631